CLINICAL TRIAL: NCT02780934
Title: Comparing Pressure Versus Simple Adhesive Dressing After Mohs Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CPHS# 29015
Record Dates: First submitted 2016-05-18; First posted 2016-05-24 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Non-melanoma Skin Cancer
Keywords: Pressure Dressing; Post-operative Care; Simple Adhesive Dressing; Mohs
MeSH Terms: interventions — Negative-Pressure Wound Therapy

ARMS (2):
- Pressure Dressing (Active Comparator): Participants randomized to this group will receive the standard post-operative dressing following their Mohs procedure: a pressure dressing consisting of high absorbency gauze and retention tape.
  Interventions: Other: Pressure Dressing
- Simple Adhesive Dressing (Experimental): Participants randomized to this group will receive the experimental post-operative dressing following their Mohs procedure: a simple adhesive dressing consisting of a non-adherent pad and transparent dressing.
  Interventions: Other: Simple Adhesive Dressing

INTERVENTIONS:
Other: Pressure Dressing — Patients in this group will receive the standard post-operative bandage: a pressure dressing consisting of high absorbency gauze and retention tape.
  Arms: Pressure Dressing
Other: Simple Adhesive Dressing — Patients in this group will receive the experimental bandage: a simple adhesive dressing consisting of a non adherent pad and transparent dressing.
  Arms: Simple Adhesive Dressing

SUMMARY:
The purpose of this study is to determine whether using a pressure- vs. simple adhesive dressing affects the postoperative course and wound healing outcomes following Mohs surgery.

DETAILED DESCRIPTION:
The investigators will randomize patients undergoing Mohs surgery to receive either a pressure or a simple adhesive dressing following their procedure. The hypothesis is that patients with the simple adhesive dressings will be more satisfied and comfortable with their wound care on follow-up. These patients are also expected to cite greater convenience managing the simple dressing at home. Finally, the investigators anticipate no difference in the number of postoperative complications between the two groups and expect that there will be a lower cost associated with the simple adhesive dressing as compared to the pressure dressing.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be considered for enrollment if they have been referred to a Mohs surgeon for consideration of Mohs surgery for non-melanoma skin cancer.

Exclusion Criteria:

* Lack of indication for Mohs
* Significant comorbidities
* Case of a high-risk location or tumor size which necessitates consultation with other specialties in advance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Assessed at the first clinical follow-up visit, 1-2 weeks following Mohs procedure
  Patients are asked to complete a survey regarding their satisfaction with their post-operative dressing. Surveys will be distributed at their first clinical follow-up visit. They are asked to rate their overall satisfaction and difficulty sleeping, bathing, and returning to normal activity following their Mohs procedure.
Complications | Assessed at the first clinical follow-up visit, 1-2 weeks following Mohs procedure
  The number of complications requiring medical attention in each arm of the study. These complications include: infection, bleeding, wound dehiscence, splitting or retained stitches, pain, and cosmetic disfigurement.